CLINICAL TRIAL: NCT00102817
Title: Somatropin (Norditropin) in Children With Growth Failure Associated With ICF Deficiency.
Brief Title: Somatropin (Norditropin) in Insulin-like Growth Factor (IGF) Deficient Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HGH-2147
Record Dates: First submitted 2005-02-01; First posted 2005-02-02 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Growth Hormone Disorder; Pituitary Dwarfism
Keywords: Growth Hormone Disorder
MeSH Terms: conditions — Dwarfism, Pituitary | interventions — Human Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: somatropin

SUMMARY:
This trial is conducted in the United States of America (USA). This is a 12 month study to determine if Norditropin is safe and effective in children with IGF deficiency.

ELIGIBILITY:
Inclusion Criteria:

* Ages 3-15
* Presence of growth failure indicated by height standard deviation score less than equal to -2
* Body mass index greater than or equal to 25th percentile for height age
* IGF concentration less than or equal to 33rd percentile

Ages: 3 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 149 (Actual)
Dates: Start 2003-05; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Change in height standard deviation score | 12 months

SECONDARY OUTCOMES:
12 months change in height standard deviation score adjusted for parent height z-score

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (26):
- United States (26):
  - Novo Nordisk Investigational Site, Los Angeles, California
  - Novo Nordisk Investigational Site, San Diego, California
  - Novo Nordisk Investigational Site, Stanford, California
  - Novo Nordisk Investigational Site, St. Petersburg, Florida
  - Novo Nordisk Investigational Site, Tallahassee, Florida
  - Novo Nordisk Investigational Site, Tampa, Florida
  - Novo Nordisk Investigational Site, Indianapolis, Indiana
  - Novo Nordisk Investigational Site, Boston, Massachusetts
  - Novo Nordisk Investigational Site, Worcester, Massachusetts
  - Novo Nordisk Investigational Site, Kalamazoo, Michigan
  - Novo Nordisk Investigational Site, Minneapolis, Minnesota
  - Novo Nordisk Investigational Site, Kansas City, Missouri
  - Novo Nordisk Investigational Site, Brooklyn, New York
  - Novo Nordisk Investigational Site, Buffalo, New York
  - Novo Nordisk Investigational Site, Rockville Centre, New York
  - Novo Nordisk Investigational Site, The Bronx, New York
  - Novo Nordisk Investigational Site, Akron, Ohio
  - Novo Nordisk Investigational Site, Cincinnati, Ohio
  - Novo Nordisk Investigational Site, Oklahoma City, Oklahoma
  - Novo Nordisk Investigational Site, Hershey, Pennsylvania
  - Novo Nordisk Investigational Site, Philadelphia, Pennsylvania
  - Novo Nordisk Investigational Site, Pittsburgh, Pennsylvania
  - Novo Nordisk Investigational Site, Columbia, South Carolina
  - Novo Nordisk Investigational Site, San Antonio, Texas
  - Novo Nordisk Investigational Site, Seattle, Washington
  - Novo Nordisk Investigational Site, Milwaukee, Wisconsin

REFERENCES:
- [Result] Cohen P, Rogol A, Kappelgaard A-M, Weng W, Germak J, Rosenfeld RG on behalf of the American Norditropin Study Group. Efficacy of IGF-I Based Growth Hormone (GH) Dose Titration in Non-GH Deficient (Non-GHD) Children with Short Stature Associated with IGF-I Deficiency (IGFD). Pediatric Academic Societies (PAS)/Lawson Wilkins Pediatric Endocrine Society (LWPES) 2007; Country: Canada City: Toronto
- [Result] Cohen P, Rosenfeld R, Rogol A, Kappelgaard A-M, Mak C, Germak J. Validation of the Efficacy and Safety of IGF-based Dose-titration in Children with Growth Failure Associated with Non-GH-deficient, IGF-I Deficiency: Results of Clinical Trial HGH 2147 on Behalf of the American Norditropin® Clinical Studies Group. 3rd International Congress of the Growth Hormone Research Society and the IGF Society 2006; Country: Japan City: Kobe
- [Derived] Cohen P, Rogol AD, Weng W, Kappelgaard AM, Rosenfeld RG, Germak J; American Norditropin Study Group. Efficacy of IGF-based growth hormone (GH) dosing in nonGH-deficient (nonGHD) short stature children with low IGF-I is not related to basal IGF-I levels. Clin Endocrinol (Oxf). 2013 Mar;78(3):405-14. doi: 10.1111/cen.12014. PMID 22924571
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com